CLINICAL TRIAL: NCT00896818
Title: The British Breast Cancer Study - National Cancer Research Network Cohort (BBC-NCRN)
Brief Title: Genes and Other Risk Factors for Second Primary Breast Cancer in Women With Breast Cancer and Their Female Family Members and Friends
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cancer Research UK (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000592728; CRUK-BBC-NCRN; UKCRN-1620; MREC--00/1/10; EU-20834
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2009-06

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Genetic Linkage; Amplified Fragment Length Polymorphism Analysis

INTERVENTIONS:
Genetic: DNA analysis
Genetic: genetic linkage analysis
Genetic: loss of heterozygosity analysis
Genetic: polymorphism analysis
Other: laboratory biomarker analysis
Other: medical chart review
Other: questionnaire administration

SUMMARY:
RATIONALE: Studying samples of blood, urine, and tumor tissue in the laboratory from patients with cancer and their female relatives and friends may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is looking at genes and other risk factors for second primary breast cancer in women with breast cancer and in their female family members and friends.

DETAILED DESCRIPTION:
OBJECTIVES:

* To identify new breast cancer susceptibility alleles in breast cancer patients and family controls.
* To compare the prevalence of known polymorphisms in genes involved in hormonal activation and degradation pathways in breast cancer patients and family controls.
* To correlate these polymorphisms with quantitative intermediate markers of susceptibility to breast cancer, such as circulating hormone levels and mammographic density.
* To perform linkage analysis to detect new susceptibility genes in larger multiple-case families combined with data on families previously collected by the Institute of Cancer Research.
* To evaluate the relationship between these polymorphisms and hormone levels in relatives and family controls.
* To compare average hormone levels in patients' unaffected first-degree relatives with family controls using urine samples from premenopausal women and urine and/or serum samples from postmenopausal women.
* To perform follow-up in a cohort of unaffected first-degree relatives at moderate-to-high risk of developing breast cancer with prospective questionnaire data and hormone measurements.

OUTLINE: Unaffected and affected first-degree female relatives and family or friend controls undergo blood sample collection once during study. Genomic DNA is purified from the blood samples for genetic analyses. Within a cohort of unaffected first-degree relatives, postmenopausal women also provide a single urine sample for hormonal assays. Hormones analyzed in the serum and/or urine of postmenopausal women include estradiol, estrone, sulphate, prolactin, androstenedione, testosterone, progesterone, 17-hydroxyprogesterone, and SHBG. Unaffected premenopausal women within the cohort provide urine samples on 6 successive days around the midpoint of their menstrual cycle and on one day towards the luteal phase of their menstrual cycle. These samples are analyzed for luteinizing hormone and metabolites of estradiol and progesterone (i.e., creatinine ratios for estrone glucuronide and pregnanediol glucuronide).

Access to case notes, mammograms, and archival tumor blocks and accompanying pathology reports of breast cancer patients and their affected relatives is requested. When tumor samples from both tumors in bilateral cases are available, these samples are analyzed to identify regions of loss of heterozygosity in which both tumors have lost the same chromosomal region.

Cancer patients and controls, including affected or unaffected first-degree relatives, relatives by marriage, or friends complete a questionnaire at baseline to provide information on demographics (i.e., personal and family), cancer diagnosis and treatment (if applicable), and known risk factors for breast cancer (i.e., lifestyle, reproductive behavior, and family history).

Study participants may be followed periodically for cancer incidence and cause-specific mortality.

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Women who have been diagnosed with contralateral or unilateral breast cancer
  * Family controls, including sisters and adult daughters of contralateral cases, female relatives by marriage
  * Unrelated controls (i.e., friends)
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Pre- or postmenopausal

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 2005-01; Primary Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of polymorphisms in candidate genes in contralateral patients and controls
Prevalence of alleles in breast cancer patients from multiple-case families and those in blood-unrelated family controls
Linkage analysis to detect new susceptibility genes in larger multiple-case families combined with data on families previously collected by the Institute of Cancer Research
Relationships between candidate gene polymorphisms and hormone levels in relatives and controls

SECONDARY OUTCOMES:
Average hormone levels in contralateral patients' first-degree relatives and controls

CONTACTS AND LOCATIONS:
Overall Officials: Julian Peto, MD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- London School of Hygiene and Tropical Medicine, London, England, United Kingdom